CLINICAL TRIAL: NCT05817812
Title: A Phase 3b Open-label Study Evaluating Physical Activity and Joint Health in Previously Treated Patients ≥12 Years With Severe Haemophilia A Treated With Recombinant Coagulation Factor VIII Fc-von Willebrand Factor-XTEN Fusion Protein (Efanesoctocog Alfa) for 24 Months
Brief Title: A Study Evaluating Physical Activity and Joint Health in Severe Haemophilia A Patients ≥12 Years Treated Once Weekly With Efanesoctocog Alfa
Acronym: FREEDOM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.BIVV001-001
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia A, Severe
Keywords: Blood coagulation disorder; Coagulation protein disorder; Haemophilia; FVIII; Efanesoctocog alfa
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Coagulation Protein Disorders | interventions — BIVV001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Efanesoctocog alfa (Experimental): All patients will be treated intravenously once weekly with 50 IU/kg efanesoctocog alfa
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — Recombinant coagulation factor VIII Fc-von Willebrand Factor-XTEN fusion protein (rFVIIIFc-VWF-XTEN)
  Other Names: BIVV001

SUMMARY:
FREEDOM is a multicentre, open-label, single-arm, phase 3b study in Europe that aims to enrol approximately 90 previously treated severe haemophilia A patients aged ≥12 years, currently on prophylaxis. After a run-in period of 30-45 days, patients will receive efanesoctocog alfa prophylaxis, 50 IU/kg once-weekly for 24 months (additional preventive dose not permitted). An activity tracker and an electronic patient diary will be used to collect data on physical activity, bleeds, factor dosing, pain, and injuries from screening throughout the study.

The primary objective is to describe changes in physical activities over 24 months on efanesoctocog alfa prophylaxis, with a primary endpoint of change from baseline in International Physical Activity Questionnaire (IPAQ) at month 24.

Secondary objectives include relationship between physical activity and other variables (bleeds, joint status, pain, injuries, and quality of life); changes in joint status as assessed by HEAD-US, HJHS and MRI; occurrence of bleeds, injuries, pain. Safety and tolerability of efanesoctocog alfa will also be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Previous treatment for haemophilia A with any marketed recombinant and/or plasma-derived FVIII for at least 150 EDs.
* Having received prophylactic treatment with any marketed recombinant and/or plasma FVIII or emicizumab per local label for at least 12 months preceding enrolment.
* Having 12 months documented pre-study treatment data regarding prophylactic treatment prescriptions and 6 months data on bleeding episodes prior to baseline visit.
* Willingness and ability to complete training in the use of the study ePD and to use the ePD in their own smartphone throughout the study.
* Willingness and ability to use the activity tracker provided by the sponsor to measure physical activity and heart rate.
* Be able and willing to administer efanesoctocog alfa intravenously at home.

Key Exclusion Criteria:

* Serious musculoskeletal and/or neurological impairment limiting the mobility and the physical ability to a degree that makes the patient unsuitable for the study as judged by the investigator.
* Other known coagulation disorder(s) in addition to haemophilia A.
* History and/or current positive inhibitor test defined as ≥0.6 BU/mL.
* Treatment with NSAIDs above the maximum dose specified in the prescribing information within 2 weeks prior to screening.
* Systematic treatment within 12 weeks prior to screening with chemotherapy and/or other immunosuppressive drugs.
* Treatment with an investigational product within 30 days or 5.5 half-lives prior to screening, whichever is longer.
* Major surgery within 12 weeks prior to screening or planned major orthopaedic surgery to occur during the study.
* At baseline visit, patients who have not been compliant in using the activity tracker.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in International Physical Activity Questionnaire (IPAQ) scoring | Baseline and month 24
  The IPAQ is a validated, 7-day recall questionnaire measuring current levels of physical activity. Scoring of the IPAQ results in a continuous variable in the form of total MET-minutes per week. Higher scores means higher physical activity level.

SECONDARY OUTCOMES:
Change from baseline in International Physical Activity Questionnaire (IPAQ) scoring | Baseline and month 12
  The IPAQ is a validated, 7-day recall questionnaire measuring current levels of physical activity. Scoring of the IPAQ results in a continuous variable in the form of total MET-minutes per week. Higher scores means higher physical activity level.
International Physical Activity Questionnaire (IPAQ) score | Baseline, month 6, 12, 18 and 24
  The IPAQ is a validated, 7-day recall questionnaire measuring current levels of physical activity. Scoring of the IPAQ results in a continuous variable in the form of total MET-minutes per week. Higher scores means higher physical activity level.
Change in mean daily minutes in physical activity | Run-in month, month 12 and 24
  Tracker-recorded
Mean daily minutes of physical activity | Per 6-month period
  Tracker-recorded
Change in type of workouts | Run-in month, month 12 and 24
  Patient and tracker reported
Change in frequency of workouts | Run-in month, month 12 and 24
  Patient and tracker reported
Change in duration of workouts | Run-in month, month 12 and 24
  Patient and tracker reported
Change in patient reported intensity of workouts | Run-in month, month 12 and 24
  The patient will report workouts in a patient diary and rate the intensity on a 5 level scale. The levels are:
  1 = easy, 2 = moderate, 3 = slightly challenging, 4 = exhausting, 5 = very exhausting.
  The changes will be calculated on a intra-patient basis
Change in tracker recorded intensity of workouts | Run-in month, month 12 and 24
  The patient will be provided with an activity tracker that will automatically record workouts when the patient is wearing the tracker. The intensity levels will be based on the heart rate and will be presented on a 4 level scale. The levels are:
  1 = out of range, 2 = fat burn, 3 = cardio, 4 = peak
Mean value of patient and tracker reported type of workouts | Per 6-month period
  Type of workout will be transcribed into a risk level of participating in a given activity for a haemophilia patient. Risk levels are based on a rating of 1-3 where level 1 represents a low risk of causing a bleeding episode and level 3 represents a high risk.
  The mean value will be calculated per 6-month period
Mean value of frequency of workouts | Per 6-month period
  Patient and tracker reported
Mean value of duration of workouts | Per 6-month period
  Patient and tracker reported
Mean value of patient reported intensity of workouts | Per 6-month period
  The patient will report workouts in a patient diary and rate the intensity on a 5 level scale. The levels are:
  1 = easy, 2 = moderate, 3 = slightly challenging, 4 = exhausting, 5 = very exhausting.
  The mean value will be calculated per 6-month period
Mean value of tracker recorded intensity of workouts | Per 6-month period
  The patient will be provided with an activity tracker that will automatically record workouts when the patient is wearing the tracker. The intensity levels will be based on the heart rate and will be presented on a 4 level scale. The levels are:
  1 = out of range, 2 = fat burn, 3 = cardio, 4 = peak
  The mean value will be calculated per 6-month period
Change in mean daily number of steps | Run-in month, month 12 and 24
  Tracker-recorded
Mean daily number of steps | Per 6-month period
  Tracker-recorded
Achieving WHO-recommended levels of MVPA | Run-in month, month 12 and 24
  Tracker-recorded
Occurrence of bleeds in relation to workouts | Baseline to month 24
Occurrence of pain in relation to workouts | Baseline to month 24
Occurrence of injuries in relation to workouts | Baseline to month 24
Occurrence of bleeding episodes impacting daily activity | Baseline to month 24
Change from baseline in Haemophilia Joint Health Score (HJHS) score | Baseline, month 6, 12, 18, 24
  The six index joints (elbows, knees and ankles) will be examined and scored. The minimum score per joint is 0, the maximum score is 20. In addition, Gait is scored on a scale from 0 to 4 based on the number of skills that are not within the normal limits.
  The total score will be the sum of scores across all six joints plus the gait score (range from 0 to 124, with 0 being normal and 124 being the most severe disease).
Change from baseline in Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) | Baseline, month 12 and 24
  The HEAD-US joint score will be calculated for six joints, the right and left ankle, knee, and elbow joints. The specific joint score is made up of three item scores, disease activity (synovitis), disease damage of articular surfaces, and disease damage of subchondral bone. Specific joint score is the sum of the three item scores for each specific joint. Its values range from 0 (minimum) to 8 (maximum).The total score represents the sum of item scores for abnormalities detected.
Change from baseline in haemophilic arthropathy assessed by the International Prophylaxis Study Group (IPSG) Magnetic Resonance Imaging (MRI) scale | Baseline, month 24
  The IPSG scale is made up of two subscores, one for soft-tissue changes and one for osteochondral changes. MRI joint score is the sum of the soft tissue and osteochondral subscores for each joint, ranging from 0-17 where 0 is absence of damage. MRI total score is the sum of joint scores across all joints.
Target joint development (three or more spontaneous bleeds into a single joint within a consecutive 6-month period) | Month 6, 12, 18, 24
  The number and proportion of patients with target joint development and the total number of target joint developed will be assessed.
Target joint resolution ( ≤2 bleeds into the joint within a consecutive 12-month period the joint is no longer considered a target joint) | Month 6, 12, 18, 24
  The number and proportion of patients with target joint resolution and the total number of target joint resolutions will be assessed
Target joint recurrence (≥3 spontaneous bleeds in a single joint within any consecutive 6-month period after target joint resolution) | Month 6, 12, 18, 24
  The number and proportion of patients with target joint recurrence and the total number of target joint recurrence will be assessed
Number of bleeding episodes | Per 6-month period and cumulative
Annualized bleeding rate (ABR) | Baseline to month 24
Total annualized efanesoctocog alfa consumption | Baseline to month 24
Number of injections and dose to treat a bleeding episode | Baseline to month 24
Pain reported via electronic patient diary | Baseline to month 24
  The patient will report pain (cause of pain, location and intensity. The intensity will reported as mild, moderately low, moderately high, severe and worst possible.
Pain intensity reported in the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale - Pain Intensity 3a | Baseline, month 6, 12, 18, 24
  The PROMIS Pain Intensity instrument assesses pain intensity on a 5-point Likert scale, ranging from 1 (had no pain) to 5 (very severe)
Pain interference reported in the Patient-Reported Outcomes Measurement Information System (PROMIS) scale - Pain interference 6a | Baseline, month 6, 12, 18, 24
  The PROMIS Pain Interference 6a is a patient-assessed instrument and is to measure pain interference on a 5-point Likert scale, ranging from 1 (not at all) to 5 (very much)
Quality of life assessed by EuroQoL 5-dimension 5-level (EQ-5D-5L) | Baseline, month 6, 12, 18, 24
  EQ-5D-5L assess 5 dimensions of health outcome (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each of the dimensions in the EQ-5D-5L questionnaire is divided into 5 levels:
  * Level 1: indicating no problem
  * Level 2: indicating slight problems
  * Level 3: indicating moderate problems
  * Level 4: indicating severe problems
  * Level 5: indicating unable to/extreme problems Patients will select a level for each dimension that best describes their health status for that dimension. A 5 digit code will be obtained, made up of the response for each dimension. This code will then be converted to an index score.The EQ-5D-5L VAS is an overall assessment of health on a scale from 1-100 that the patient provides at the end of the EQ-5D-5L questionnaire. 100 represents the best health you can imagine and 0 represents the worst health you can imagine.
Assessment of treatment preference | 24 months
  This will be assessed with the Treatment Preference Survey that consists of 2 questions on perceived impact of treatment.
The occurrence of adverse events and serious adverse events | From screening to month 24
The occurrence of clinically significant changes | Baseline, month 6, 12, 18, 24
  Assessed by physical examination, vital signs and laboratory tests
Development of inhibitors (neutralizing antibodies directed against FVIII) | Baseline, month 6, 12, 18, 24
  Determined via the Nijmegen modified Bethesda assay
The occurrence of thrombotic and embolic events | From screening to month 24
Number of non-study medical care encounters | From baseline to month 24
  The number and proportion of patients having non-study medical care encounter visits will be described, as well as the corresponding total number of visits.
Duration of non-study medical care encounters | From baseline to month 24
  The duration of non-study medical care encounter visits will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, MD, PhD, Study Director — Swedish Orphan Biovitrum AB
Locations (30):
- Investigational Site, Vienna, Austria
- Investigational Site, Zagreb, Croatia
- Czechia (2):
  - Investigational Site, Brno
  - Investigational Site, Prague
- France (4):
  - Investigational Site, Bordeaux
  - Investigational Site, Le Kremlin-Bicêtre
  - Investigational Site, Marseille
  - Investigational Site, Strasbourg
- Germany (4):
  - Investigational Site, Berlin
  - Investigational Site, Frankfurt
  - Investigational Site, Giessen
  - Investigational Site, Hamburg
- Investigational Site, Athens, Greece
- Investigational Site, Dublin, Ireland
- Italy (5):
  - Investigational Site, Catanzaro
  - Investigational Site, Florence
  - Investigational Site, Naples
  - Investigational Site, Parma
  - Investigational Site, Rome
- Investigational Site, Utrecht, Netherlands
- Investigational Site, Oslo, Norway
- Investigational Site, Ljubljana, Slovenia
- Spain (3):
  - Investigational Site, Barcelona
  - Investigational Site, Madrid
  - Investigational Site, Oviedo
- Sweden (2):
  - Investigational Site, Lund
  - Investigational Site, Solna
- United Kingdom (3):
  - Investigational Site, Canterbury
  - Investigational Site, Newcastle upon Tyne
  - Investigational Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sobi's data sharing criteria and process for requesting access can be found at: https://www.sobi.com/en/policies
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: https://www.sobi.com/en/policies